CLINICAL TRIAL: NCT01709526
Title: Prospective Study the Adolescent Inpatients Rehabilitation
Brief Title: How the Adolescent Inpatients Are Rehabilitated After Discharge
Acronym: AdolInpRehabi
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study couldn´t start due to investigator
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Helena Pehkonen, assistant, Kuopio University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUH5702803; KUH5702803
Record Dates: First submitted 2011-06-29; First posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Psychiatric Diseases
Keywords: Psychosocial functioning; Cognitive performance of inpatients; Psychiatric diseases
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Improvement after psychiatric inpatient treatment (Other)
  Interventions: Behavioral: Improvement after psychiatric inpatient treatment

INTERVENTIONS:
Behavioral: Improvement after psychiatric inpatient treatment — Cognition, psychosocial functioning
  Other Names: After adolescents treatment

SUMMARY:
The aims of this six month follow-up study are which treatment components will correlate or which clinical treatments interventions contribute adolescent inpatients recovering in the psychiatric treatment after discharge. Comparisons will be made between the 47 adolescents aged 13 to 18 years, with major depression and conduct disorders, and between those with and without suicide attempts by multivariate analyses. Are the adolescent psychiatric inpatients recovered?

DETAILED DESCRIPTION:
The whole prospective study sample consisted of 63 adolescents aged 13 to 18 years (40 girls and 23 boys)referred for psychiatric treatment to the adolescent psychiatric inpatient unit of Kuopio University Hospital, Finland. This study is part of the "Kliininen Laatuprojekti"- Depression Project in Kuopio University Hospital. Researcher UH, Doctor of Philosophy, has been the head of the study project. She has done this study by carrying, analysing, doing articles and writing abstracts and keeping lectures and congress sessions in Finland and aboard. In the same time she has done clinical work by caring adolescents in the hospital ward and in the therapy settings. UH has been the first writer in the articles, one article in national and three in international articles. This Doctoral dissertation has been presented 17th November 2007, supervisor was professor, MD. Mauri Marttunen.

The prospective study set out to investigate gender differences, psychosocial and cognitive functioning, self-image, and changes in these structured parameters, and the role of working alliance. More girls than boys were admitted to inpatient care. Mood and conduct disorders were the most common diagnoses. Girls more commonly had poor family relationships but more peers than boys. Violent and destructive behaviour were more common among boys, and they performed worse in tests assessing nonverbal cognitive performance and total immediate recall memory than girls. Both girls and boys had an impaired IQ at entry. Major impairment in functioning in several areas such as school, family relations, judgement and thinking was found among both genders.

The psychosocial functioning and cognitive performance of inpatients improved during treatment.

There were also improvements in intrapsychic constructs: in the psychological self-image, especially body-image, and in relationships with family members, particularly among emotionally-disturbed adolescents. Cognitive performance was significantly enhanced among subjects both with a good and with a poor working alliance. According to multivariate analyses, a better quality of working alliance and a greater number of therapy sessions were associated with positive changes in cognitive performance and self-image.

When subjects with major depression and conduct disorder were compared, nonverbal cognitive and general cognitive performance, body and self-image, and overall psychosocial functioning improved in both groups of subjects during treatment. More positive changes in self-image and family functioning were found among subjects with MDD.

Suicidal adolescents' treatment compliance and outcome were as good as those of non-suicidal patients. Their psychosocial functioning, cognitive performance, and both the psychological self and body-image improved during treatment. Positive changes in body-image associated significantly with a higher probability of improvement in psychosocial functioning, while a higher GAS score at entry was associated with a lower probability of functional improvement. In clinical practice, attention needs to be paid to structured assessment of adolescent psychiatric inpatients. This study suggests a need to combine at least regular individual therapy, pharmacotherapy, family interventions, and a school program. Since a good working alliance between the therapist and the adolescent patient seems to modify the treatment outcome, particular attention to creating a good alliance with the patient and intensive involvement of the parents in treatment are recommended. Prospective studies with a sufficient follow-up after discharge and well-designed intervention studies among adolescent inpatients are needed.

Now it is interested in how they are in recovery with the role of working alliance and improvement in the psychosocial functioning after discharge?

ELIGIBILITY:
Inclusion Criteria:

* psychiatric disease
* adolescents
* inpatient treatment

Exclusion Criteria:

* emergency psychiatric treatment
* under 4 weeks treatment

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2009-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Hintikka, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland